CLINICAL TRIAL: NCT00311701
Title: A Retrospective Chart Review to Assess the Safety of Oseltamivir (Tamiflu®) Compared to Alternate Antiviral Therapy (Amantadine or Rimantadine) Administered to Children Less Than 12 Months of Age With Diagnosed or Suspected Influenza (CASG 113)
Brief Title: Chart Review of Antivirals for Influenza in Infants
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Other Study IDs: 05-0111; CASG 113; N01AI30025C; N01AI30025 (NIH)
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2007-10

CONDITIONS: Influenza
Keywords: Influenza, pediatric
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This retrospective study conducted in Canada and the US involves a chart review to assess the safety of oseltamivir (Tamiflu®) compared to alternate antiviral therapy, amantidine or rimantidine, administered to children less than 12 months of age with diagnosed or suspected influenza. The objectives are to describe the frequency of neurological and all other adverse events possibly related to administration of these antivirals in these infants. Investigators will also compare frequency of adverse events at various doses of oseltamivir in these children. Critical endpoints to be collected include frequency and severity of adverse events, particularly those relating to central nervous system complications. A sub-investigator will travel to each of the participating sites to collect data related to each infant's health prior to becoming ill, health status at time of influenza diagnosis, dosing regimen, reported neurological events post-dosing, and all reported adverse events post-dosing.

DETAILED DESCRIPTION:
The study is a retrospective review of charts of children less than 12 months of age that were diagnosed with influenza and treated with oseltamivir. The chart review will focus on assessment of neurological and other adverse events that may have been related to the administration of oseltamivir. A control population will consist of children less than 12 months treated with either rimantadine or amantadine. The administration of oseltamivir to children at high risk (i.e. immunocompromised hosts) less than 12 months old with influenza is frequently considered in medical practice despite the findings of neurotoxicity in a juvenile rat study. Since oseltamivir is the only active treatment against H5N1 influenza strains, it is imperative to understand the ramifications of its potential widespread use in very young infants in the event of an outbreak. This study is designed to gather documented evidence by which the circumstances of use and defined outcomes can be described. Patient selection will be made by review of hospital inpatient medical records, emergency room medical records and/or pharmacy records to identify patients less than 1 yr old dosed with oseltamivir suspension. Redacting the charts will be done in a manner that will obscure personal health information (individual identifiers) without obscuring the necessary clinical data. A separate research data collection form will be prepared on which critical information can be transcribed that would subsequently be available for analysis. Critical information to be captured at the time of initiating oseltamivir treatment includes: age, birth history, gender, underlying medical conditions, presenting influenza symptoms, if done, type of flu test and dose regime. Critical endpoints to be collected will include the frequency and severity of adverse events, particularly those relating to central nervous system complications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female study participants less than 12 months of age
2. Suspected or laboratory diagnosis of influenza
3. Treated with oseltamivir, rimantadine or amantadine

Exclusion Criteria:

None listed

Max Age: 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2005-11; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Locations (16):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Pulaski, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital and Health Center, San Diego, California
  - University of Colorado, Denver, Colorado
  - Washington University in St. Louis, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - MetroHealth Medical Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- University of Alberta, Edmonton, Alberta, Canada